CLINICAL TRIAL: NCT06964386
Title: Effect of Specially Designed Balance Board on Standing Balance in Children With Diplegic Cererbral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Zeinab Mohamed Hassan Ewida, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Zeinab-004238
Record Dates: First submitted 2025-05-01; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Balance Board; Standing Balance; Diplegic Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the traditional program (Experimental): twenty Children in group A received designed physical therapy program in addition to traditional balance training
  Interventions: Other: The traditional physical therapy rehabilitation exercises; Other: balance training on traditional balance board
- balance training exercises (Active Comparator): twenty Children in group B received the same designed physical therapy program in addition to balance training exercises on special form of balance board
  Interventions: Other: The traditional physical therapy rehabilitation exercises; Other: program on special form of balance board

INTERVENTIONS:
Other: The traditional physical therapy rehabilitation exercises — It included 30 minutes of exercises as:
  * Incorporated stretching (adductors, calf, and hamstring muscles)
  * Range of motion for hip, knee, and ankle joints.
  * Core stability exercises.
  * climbing stairs and weight-bearing activities for strengthening, such as sit-to-stand and attaining standing position by half kneeling
Other: balance training on traditional balance board — Balance training included: - Side stepping - Stepping backward - Changing the center of gravity in one-foot balance.
  Arms: the traditional program
Other: program on special form of balance board — Standing holding on the sticks of balance board (first by two sticks, then graduated by one stick).
  2- Changing the grasp of hand on sticks (reciprocal catching the sticks by right and left hand).
  3- Stride standing on balance board. 4- Make exercises advanced by remove sticks and throwing the ball. 5- All previous exercises do with eye closed and eye opened
  Arms: balance training exercises

SUMMARY:
This was done to:

1. To determine the effect of a specially designed balance board on balance ability.
2. To determine the effect of the traditional balance training program on balance ability.
3. To compare between the effect of a specially designed balance board and the traditional balance training program on balance ability.

DETAILED DESCRIPTION:
Children with cerebral palsy (CP) often experience abnormal posture, loss of motor control, and poor trunk control, leading to limitations in daily activities. Improving balance abilities is crucial for maintaining equilibrium in sensory environments. Vestibular stimulation can help develop feed-forward mechanisms and new functional skills. This study aims to improve balance abilities in children with diplegic CP, explore the impact of balance boards on vestibular and hand function, and assist mothers in their child's improvement.

ELIGIBILITY:
Inclusion Criteria:

1. Their ages ranged from 4 to 8 years old.
2. The degree of spasticity ranged from grade 1 or 1+ according to Modified Ashworth Scale
3. They were at level I or II on gross motor function classification scale.
4. They were able to follow verbal command or instructions.

Exclusion Criteria:

Children were excluded if they had one of the following :

1. Fixed deformities of lower limbs.
2. Visual or auditory problems.
3. History of surgical interference in lower limbs less than six months.
4. Botulinum toxin injections to the lower limb during the previous 4 months.
5. Mental retardation.
6. Fixed deformity

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
assessment of degree of spasticity | at baseline and after 3 months
  Assessment of tone involves the clinician passively moving the patient's joints slowly and quickly and rating the degree of resistance felt to rapid stretch, typically as increased or decreased relative to a presumed normal (Hugos and Cameron, 2019). Only spastic diplegic children with grade 1 and 1+ will be included in the study

SECONDARY OUTCOMES:
Assessment of change of gross motor function level | at baseline and after 3 months
  This study will involve children with diplegic cerebral palsy at level II, who can walk, climb stairs, and perform gross motor skills like running and jumping. They will be allowed to engage in functional activities without interruption from caregivers or therapists. The study will record their activities using gross motor function classification system, taking about 10 minutes. Children with level II may struggle with long distances, balancing, and uneven terrain, and may require assistance with physical assistance or wheeled mobility.
assessment of change of balance | at baseline and after 3 months
  it is an electronic balance board with HUMAC software on a laptop. Calibration was performed according to manufacturer guidelines. Participants stood with hands by their sides, without assisted devices. A sight target was taped to the wall. Participants stood quietly for one minute before testing.
assessment of change of pediatric balance | at baseline and after 3 months
  The pediatric balance scale is a tool designed for children and adolescents aged five to 15 years to assess their static and dynamic balance. It consists of 14 items with scores ranging from 0 to 4, with a maximum score of 56. The scale has test-retest and interrater reliability of 0.998 and 0.997 in school-aged children with mild to moderate motor impairment. It requires minimal specialized equipment, such as an adjustable seat, chair, stopwatch, footrest, eraser, tape measure, and child-sized foot molds.

CONTACTS AND LOCATIONS:
Locations (1):
- out-patient clinic, faculty of physical therapy, Cairo university, Cairo, Egypt